CLINICAL TRIAL: NCT01091727
Title: Prospective Randomized Double-blind Trial of Intravesical Injection of Botulinum Toxin A Versus Saline for Neurogenic Detrusor Overactivity and Urinary Incontinence Related to Spinal Cord Injury or Multiple Sclerosis
Brief Title: Intravesical Injection of Botulinum Toxin A Versus Saline for Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sender Herschorn, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0922006
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Neurogenic Detrusor Overactivity
Keywords: Neurogenic; Detrusor; Overactive; Overactivity; Bladder; Spinal; Cord; Injury
MeSH Terms: conditions — Cone-Rod Dystrophies; Wounds and Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin A (Experimental): Botulinum toxin A 300U diluted with sterile saline (1 ml per injection site) and injected into 30 sites of the bladder, sparing the trigone.
  Interventions: Drug: Botulinum toxin A
- Placebo (Placebo Comparator): Sterile saline 30 cc injected into 30 sites in the bladder, sparing the trigone.
  Interventions: Drug: Botulinum toxin A

INTERVENTIONS:
Drug: Botulinum toxin A — Comparison of intra-detrusor injection of 300U of Botulinum toxin A versus placebo for effect on neurogenic detrusor overactivity and urinary incontinence.
  Other Names: Botox

SUMMARY:
This is a prospective, multicentre (7 sites), randomized, double-blind, study comparing intravesical injection of BOTOX to placebo in 56 subjects with NDO secondary to spinal cord injury or multiple sclerosis. Study subjects will be randomized to one of the following two treatment groups:

Group 1 n=28 BOTOX - 300U Group 2 n=28 Placebo BOTOX (saline)

All study subjects will receive one injection cycle (BOTOX 300U or Placebo) at Visit 2 (Treatment, Day 0) as per Supplement III. The study duration is approximately 61 weeks and consists of a Pre-Treatment Evaluation, a Treatment/Randomization Visit (Visit 2, Day 0), Telephone Follow-ups at 1, 3 and 4 weeks post-treatment, and Follow-up Visits at 6, 24 and 36 weeks (Visits 3 to 5). At Week 36, subjects will be offered open-label BOTOX 300U and will be followed for an additional 6 months, returning for evaluations at Weeks 48 and 60.

DETAILED DESCRIPTION:
This is a prospective, multicentre (7 sites), randomized, double-blind, study comparing intravesical injection of BOTOX to placebo in 56 subjects with NDO secondary to spinal cord injury or multiple sclerosis. Study subjects will be randomized to one of the following two treatment groups:

Group 1 n=28 BOTOX - 300U Group 2 n=28 Placebo BOTOX (saline) All study subjects will receive one injection cycle (BOTOX 300U or Placebo) at Visit 2 (Treatment, Day 0) as per Supplement III. The study duration is approximately 61 weeks and consists of a Pre-Treatment Evaluation, a Treatment/Randomization Visit (Visit 2, Day 0), Telephone Follow-ups at 1, 3 and 4 weeks post-treatment, and Follow-up Visits at 6, 24 and 36 weeks (Visits 3 to 5). At Week 36, subjects will be offered open-label BOTOX 300U and will be followed for an additional 6 months, returning for evaluations at Weeks 48 and 60.

ELIGIBILITY:
Inclusion Criteria

1. Outpatient, male or female subjects, of any race, between 18 and 75 years of age. Female subjects of childbearing potential must have a negative urine pregnancy test result on the day of Treatment (Visit 2) and practice a reliable method of contraception.
2. Subjects with a neurogenic bladder and detrusor overactivity secondary to either a spinal cord injury or multiple sclerosis.
3. Subjects with urinary incontinence (minimum of one occurrence per day) despite current treatment.
4. Subjects with serum creatinine within normal limits and normal renal function.
5. Subjects on a stable dose (minimum one month) of concomitant medication for NDO.
6. Subjects able to understand the requirements of the study, including completing questionnaires and signing Informed Consent.

Exclusion Criteria

1. Female subjects who are pregnant (positive urine pregnancy test), are planning to become pregnant during the study period, have an infant they are breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
2. Subjects with a history of transurethral sphincterotomy, bladder neck or prostatic resection, previous bladder surgery including myomectomy or augmentation cystoplasty.
3. Subjects with chronic indwelling catheters.
4. Subjects with any medical condition that may increase their risk of exposure to botulinum toxin including diagnosed Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis or any other disease that might interfere with neuromuscular function.
5. Subjects with an allergy or sensitivity to any component of BOTOX® (Section 5.2).
6. Subjects unable to discontinue any agents that might interfere with neuromuscular function (i.e., aminoglycoside antibiotics, curare-like agents, etc.).
7. Subjects with, in the opinion of the Investigator, unstable stable multiple sclerosis.
8. Subjects with known, uncontrolled systemic disease.
9. Subjects with evidence of recent alcohol/drug abuse.
10. Subjects who, in the opinion of the Investigator, have a significant condition or situation that may put the subject at significant risk, confound the study results, or interfere significantly with the subject's participation in the study.
11. Subjects with a history of poor cooperation, non-compliance, or unreliability.
12. Subjects currently participating in an investigational drug study or who have participated in an investigational drug study within 30 days of the Baseline Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy | 36 weeks
  Frequency of Incontinence Episodes over 3 days (3-Day Voiding Diary)

SECONDARY OUTCOMES:
Efficacy | 36 weeks
  Maximum Detrusor Pressure During Filling;Volume at Maximum Detrusor Pressure During Filling at 6 Wks;Volume at Maximum Detrusor Pressure During Filling other than at 6 Wks;Reflex Detrusor Volume at First Contraction; Maximal Bladder Capacity;Frequency of micturition; Bladder Compliance;ICIQ,DBICI,I-QOL Incontinence intervals, number of pads used, amount leaked, degree of urgency Intermittent Catheterizations;Urine volume obtained during catheterization Timing and reduction or cessation of anticholinergic medication

CONTACTS AND LOCATIONS:
Overall Officials: Sender Herschorn, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada